CLINICAL TRIAL: NCT05947903
Title: Validation of the European Oncology Quality of Life Toolkit. A European Pilot Survey.
Brief Title: Validation of the European Oncology Quality of Life Toolkit
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other); German Cancer Research Center (Other); Oslo University Hospital (Other); The Netherlands Cancer Institute (Other); Hospital del Mar Research Institute (Unknown); Istituto Europeo di Oncologia (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); UNICANCER (Other); EAPC (Unknown); Institut Curie (Other); EUROPEAN CANCER ORGANISATION (Unknown); DIGICORE/IFO (Unknown); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Alleanza Contro il Cancro (Other); Istituti Fisioterapici Ospitalieri (Other); STICHTING NEDERLANDS INSTITUUT VOOR ONDERZOEK VAN DE GEZONDHEIDSZORG (Unknown); University of Milan (Other); SporeData OÜ (Unknown); ORGANISATION OF EUROPEAN CANCER INSTITUTES (Unknown); FEDERAZIONE ITALIANA DELLE ASSOCIAZIONI DI VOLONTARIATO IN ONCOLOGIA (Unknown); Medical University Innsbruck (Other); SDRUZHENIE ASOTSIATSIA NA PATSIENTITE SONKOLOGICHNI ZABOLYAVANIA I PRIYATELI (Unknown); FEDERATIA ASOCIATIILOR BOLNAVILOR DE CANCER (Unknown); University of Leeds (Other); The Leeds Teaching Hospitals NHS Trust (Other); Region Hovedstaden (Bispebjerg Hospital & Rigshospitalet) (Unknown)
Responsible Party: Sponsor
Other Study IDs: INT 106/23
Record Dates: First submitted 2023-06-28; First posted 2023-07-17 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Survivorship; Palliative Care
Keywords: Quality of life; cancer; questionnaire; validation; survivorship; palliative care; Patient Reported Outcomes
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A) EUonQoL-Kit - Active Treatment module: EUonQoL-Kit questionnaire specifically designed and administered to patients undergoing/having recently completed curative treatment for early-stage cancers OR undergoing/having recently completed non-curative treatment for advanced or metastatic cancers, including disease controlling/life prolonging tumour-directed treatment.
  Interventions: Other: Administration of the EUonQoL-Kit - Active Treatment questionnaire
- B) EUonQoL-Kit - Survivors module: EUonQoL-Kit questionnaire specifically designed and administered to people being disease-free without evidence of active cancer, and at least one year off active treatment (with the exception of long-term adjuvant hormonotherapy).
  Interventions: Other: Administration of the EUonQoL-Kit - Survivors questionnaire
- C) EUonQoL-Kit - Palliative Care module: EUonQoL-Kit questionnaire specifically designed and administered to patients with advanced cancers with projected prognosis <12 months and Eastern Cooperative Oncology Group (ECOG) ≥2 OR referred to a specialist palliative care team for symptom control, OR receiving non-curative systemic treatment or radiotherapy purely for symptom control.
  Interventions: Other: Administration of the EUonQoL-Kit - Palliative Care questionnaire

INTERVENTIONS:
Other: Administration of the EUonQoL-Kit - Active Treatment questionnaire — Electronic questionnaire to be administered to patients in active treatment.
  Groups: A) EUonQoL-Kit - Active Treatment module
Other: Administration of the EUonQoL-Kit - Survivors questionnaire — Electronic questionnaire to be administered to cancer survivors.
  Groups: B) EUonQoL-Kit - Survivors module
Other: Administration of the EUonQoL-Kit - Palliative Care questionnaire — Electronic questionnaire to be administered to patients in palliative care.
  Groups: C) EUonQoL-Kit - Palliative Care module

SUMMARY:
The improvement or preservation of quality of life (QoL) is one of the three pillars of the European Union (EU) Mission on Cancer, which underpins the needs of patients from cancer diagnosis throughout treatment, survivorship, and advanced terminal stages. Clinical studies and real-world data show that the use of Patient Reported Outcome Measures (PROMs) for QoL assessment in routine oncology practice has positive effects on patient wellbeing and healthcare resource utilization. However, full implementation of PROMs is not yet part of standard of care and is not adequately considered in cancer policies and programs.

A comprehensive tool incorporating the perspective of patients at different stages of the disease trajectory and widely applicable across Europe is still lacking.

The European Oncology Quality of Life Toolkit (EUonQoL-Kit) is a unified patient-centred tool for the assessment of QoL, developed from preferences and priorities of people with past or current cancer experience. The EUonQoL-Kit includes three electronic questionnaires, specifically designed for different disease phases (patients in active treatment, survivors, and patients in palliative care), available in both static and dynamic (Computer Adaptive Testing, CAT) versions and in several European languages.

This is a multicentre observational study, with the following aims:

* The primary aim is to perform the psychometric validation of the EUonQoL-Kit.
* Secondary aims are to assess its acceptability, to validate the static and dynamic versions against each other, and to provide estimates of QoL across European countries.

The EUonQoL-Kit will be administered to a sample of patients from 45 European cancer centres. The sample will include patients in active treatment (group A), survivors (group B), and patients in Palliative Care (group C).

Each centre will recruit 100 patients (40 from group A, 30 from group B, 30 from group C), for an overall sample size of 4,500 patients (at least 4,000 patients are assumed to be enrolled, due to an expected lower recruitment rate of 10-15%). Three sub-samples of patients (each corresponding to 10% of the total sample for each centre) will fill in an additional questionnaire:

* FACT-G (Functional Assessment of Cancer Therapy - General) and EQ-5D-5L (5-level European Quality of Life Five Dimension), to test concurrent validity.
* Live-CAT version, to validate the static and dynamic versions against each other.
* EUonQoL-Kit, at least 1 hour after the first completion, to assess test-retest reliability.

DETAILED DESCRIPTION:
Several patient-reported questionnaires have been developed and validated to measure quality of life (QoL) of cancer patients. However, a comprehensive tool, developed in close collaboration with people who have experienced cancer, widely applicable across Europe and tailored to the health status of the individual patient, is lacking. Such a tool will be important for incorporating the patient's perspective into the evaluation of policies and programs addressing cancer at the European level.

The European Oncology Quality of Life Toolkit (EUonQoL-Kit) is a unified patient-centred tool for the assessment of QoL based on preferences of cancer patients and survivors. It is developed from a patient perspective, administered digitally, available in the languages of the European Union (EU) 27 and several associated countries, and applicable in future surveys to contribute to the EU's mission on cancer. It includes three static questionnaires specifically developed for different disease phases (patients in active treatment, survivors, and patients in palliative care), and three dynamic versions of the same questionnaires based on Item Response Theory (IRT) and Computer Adaptive Testing (CAT).

This is an observational study aimed to perform the psychometric validation of the EUonQoL-Kit through its first large scale application in a pan European pilot survey.

The EUonQoL-Kit will be tested in a sample of cancer patients and survivors from 45 oncological centres located in 33 European countries. The sample will include patients in active treatment (group A), survivors (group B), and patients in Palliative Care (group C). Each centre will recruit a sample of 100 participants (40 from group A, 30 from group B, 30 from group C), stratified for primary diagnosis: lung cancer, breast cancer, colorectal cancer, haematological malignancies, prostate cancer, others.

In each centre, data collection will be performed in pre-identified outpatient clinics and inpatient wards. Participation in the study will be offered to eligible patients until the pre-defined sample size is reached.

All patients in the sample will fill in the EUonQoL-Kit. Additionally, three subgroups of patients will be proposed to fill in the following additional questionnaires:

* FACT-G and EQ-5D-5L, to evaluate concurrent validity ("concurrent validity" sub-sample: 10% of the overall sample, stratified for the three disease conditions: A, B, and C).
* Live CAT version of the EUonQoL-Kit, to validate the static and dynamic versions against each other ("live CAT" sub-sample: 10% of the overall sample, stratified for the three disease conditions).
* EUonQoL-Kit, a second time, (at least 1 hour after the first administration), to assess test-retest reliability ("test-retest" sub-sample: 10% of the overall sample, stratified for the three disease conditions).

The development of the EUonQoL-Kit has involved multiple stakeholder groups, also including patients, through different steps:

* Systematic search, collection, and analysis of existing validated QoL tools, metrics, item banks in databases to identify QoL dimensions not adequately covered by existing tools.
* A mixed-method study including patient interviews, a Delphi survey with patients and healthcare providers, aimed at collecting patient priorities and preferences on QoL dimensions, followed by a usability testing of a preliminary version of the EUonQoL-Kit.
* Development of the EUonQoL-Kit, including three static questionnaires specifically developed for patients in active treatment, survivors and in palliative care, and three dynamic versions of the same questionnaires. The final version of the six questionnaires will be submitted as an amendment to the current protocol when available.
* Translation and cultural adaptation of the EUonQoL-Kit across European countries.

The CAT version of the EUonQoL-Kit requires an item bank containing IRT-calibrated items (questions) and an algorithm for selecting the most relevant item to ask, based on the previous answers. Such dynamic system ensures that each patient is asked the most relevant and informative items.

CAT/IRT-based technology will be implemented as:

* Short forms within the EUonQoL-Kit static version. Three static versions will be designed to secure the optimal fit between items and patient groups.
* Live CAT, within the EUonQoL-Kit dynamic version. Each item is selected based on the previous answers, while the patient completes the questionnaire.

The final EUonQoL-kit will include both traditional and CAT/IRT-based items.

The overall sample size is planned to be 4,500 patients. Expecting a lower recruitment rate of 10-15%, at least 4,000 patients will be enrolled, a number suitable for data analyses.

Scientifically sound recommendations on statistical power/sample size in validation studies are lacking and minimum rule-of-thumb requirements are provided. The highest number of participants recommended for exploratory and confirmatory factor analyses (EFA & CFA) is 1,000; thus, the sample size by subgroup mentioned above is appropriate to evaluate construct validity.

Analyses of the primary aim will include:

* EFA & CFA to assess structural validity. The sample will be divided into two random sub-samples, stratified by disease stage and country. The first sub-sample will be used to perform EFA, and the model obtained will be confirmed by CFA in the second sub-sample. Goodness-of-fit will be measured by the Root Mean Square Error of Approximation, Comparative Fit Index, and Tucker-Lewis Index.
* Distribution of scale scores, examined by calculating the observed range, floor and ceiling effects, and statistics of central tendency and dispersion.
* Reliability in terms of internal consistency (estimated with Cronbach's alpha coefficient of multi-item scales) and reproducibility (agreement between the two administrations of EUonQoL-Kit estimated with the Intra-class Correlation Coefficient).
* Concurrent validity, assessed by the multi-trait multimethod matrix between the EUonQoL-Kit and the FACT-G/EQ-5D-5L questionnaires.
* Construct validity based on hypotheses-testing, assessed through the patterns of EUonQoL-Kit scores across known groups defined by variables such as disease stage, treatment, and Eastern Cooperative Oncology Group performance status. Mean differences among groups will be tested with ANOVA, and the magnitude of the difference between them will be estimated by Effect Size coefficient: > 0.8 high, 0.5 moderate, and 0.2 low.
* Test of Differential Item Functioning, used to assess item equivalence.

Analyses of the secondary aims will include:

* Assessment of acceptability and respondent burden, based on the response rate and percentage of missing items, as well as the time needed to complete the questionnaire.
* Validation of the static and dynamic versions of the EUonQoL-Kit against each other, performed by 1) comparing scores obtained with the static and dynamic versions to test if they produce interchangeable results; and 2) assessing whether the items selected for the static versions should be adjusted to obtain optimal assessment.
* To analyse QoL inequalities across clusters of populations, countries, and healthcare systems, multi-level regression models will be applied across three levels: individual, cancer centre and country. It will also be explored whether the magnitude of subgroup differences (e.g., for age or education) varies across countries.
* Analysis of QoL disparities across different patient groups will include gender, ethnicity, religion, geographical area, psychological and socio-economic factors, and education level.

Data collected include personal information belonging to special categories, like health-related data, origins, lifestyles etc. Legal basis to collect and process information is the data subject consent, which is necessary to take part in this study. A data protection expert will assess the impact on data protection throughout the duration of the study. Patient registration and CRF data collection will be centralized through the CRF.net platform, developed and owned by Istituto Nazionale Tumori, IRCCS - Fondazione G. Pascale, Napoli (INT-NA) and released with the GPL v3 license. Data will be stored by INT-NA on cloud services provided by Telecom Italia S.p.A. and located in Acilia (Italy).

Patient-reported data associated to QR codes will be collected by an ad hoc mobile app developed by Clinical Research Technology (CRT), Salerno (Italy).

The CAT version of EUonQoL-Kit will be administered through the integration of a CAT engine provided by the European Organization for Research and Treatment of Cancer (EORTC), sited in Bruxelles (Belgium).

Data processing is managed by:

* Istituto Nazionale Tumori, IRCCS - Milan (INT): INT serves as the data controller.
* Istituto Nazionale Tumori, IRCCS - Fondazione G. Pascale, Napoli (INT-NA). INT-NA will be appointed as data processor under article 28 GDPR and will be responsible for patient enrolment, questionnaire assignment through the generation of a QR code, clinician reported data collection through the electronic Case Report Form (eCRF), management of the interface with the CAT engine and with the mobile app for the administration of EUonQoL-kit items.
* CRT: based on a QR code provided by CRF.net platform, the mobile app administers specific QoL questionnaires for specific subgroup of patients. For each item administered, the app will directly transfer the answer to the platform, without recording/storing any content. Such a procedure avoids any possibility to link contents to patients' IDs.
* EORTC: in case of the dynamic EUonQoL-Kit administration, EORTC CAT will be appointed as data processor under article 28 GDPR and will get access to each pseudonymized answer as provided by the CRF.net platform. The EORTC CAT will delete any content once the questionnaire has been submitted including scores sent to the CRF.net platform.

The CRF.net platform is accessible online by investigators and data managers through username and password and is protected through encrypted data certified by SSL certificates and HTTPS protocols. For each registered patient, the CRF.net platform generates a Quick Response (QR) code that will be scanned with the tablet to allow the patient to complete the questionnaires.

The interface of the platforms allows data review and cleaning in the central archive directly (with a limited and controlled access of data-managers and investigators). Each operation done in the archive database is registered through track-change.

Each participating centre will receive tablet devices from the sponsor to get access to the CRF.net platform and collect data directly from patients. Results will be shared as open data in a completely anonymous and aggregated form. After 5 years since data collection, all personal information related to the study, including informed consents, will be anonymized/destroyed according to the delay stated by the Ethics Code on data processing for statistics or scientific research purposes issued by the Italian Data Protection Authority under article 20, par. 4, LD 101/2018.

Patients could exercise their rights by submitting requests to the staff identified in the private information. All centres have appointed a data protection officer under the General Data Protection Regulation (GDPR) and an internal data breach policy.

This study was designed and shall be implemented and reported in accordance with national and European legal and ethical requirements. Moreover, the survey will follow the ethical principles laid down in the Declaration of Helsinki and the ethical principles of observational research on potentially fragile patients.

The protocol, Informative Sheet, and Informed Consent Form must be reviewed and approved by ethics committees of each centre involved. No study procedure can be performed before the written informed consent has been provided.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more.
* Present or past histologically confirmed diagnosis of solid tumour or haematological malignancy.
* Being in one of these three conditions: A) Patients in active treatment; B) Survivors; C) in Palliative Care.
* Native tongue or fluent in the language of the questionnaire
* Written informed consent to the study.

Exclusion Criteria:

* Cognitive impairment preventing the completion of the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in one of the following three conditions will be screened for their eligibility:
  A) In active treatment: Undergoing or recently completed curative treatment for early-stage cancers OR undergoing or recently completed non-curative treatment for ad-vanced or metastatic cancers, including disease controlling/life prolonging tumour-directed treatment.
  B) Survivors: Being disease-free without evidence of active cancer, and at least one year off active treatment (with the exception of long-term adjuvant hormonotherapy).
  C) Palliative Care (PC): patients with advanced cancers with projected prognosis <12 months and ECOG ≥2 OR referred to a specialist palliative care team for symptom control.
  OR receiving non-curative systemic treatment or radiotherapy purely for symptom control.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability of the EUonQoL-Kit static version | All assessments at time of administration of the questionnaires, apart reproducibility that will be assessed with a re-test at least after 1 hour for all patients
  Exploratory and confirmatory factor analyses, distribution of the scales' scores, reliability in terms of internal consistency and reproducibility, concurrent and construct validity, differential item functioning.

SECONDARY OUTCOMES:
Acceptability of the EUonQoL-Kit | At day 1
  Acceptability of the EUonQoL-Kit and reasons for refusal, including patient burden in filling in the questionnaire
Validation of the EUonQoL-Kit dynamic (CAT) version | At day 1
  Comparison of the scores obtained with the static and dynamic versions to test if they produce similar, interchangeable results; assessment to test whether the items selected for the static version and the related CAT-settings should be adjusted to obtain optimal assessment.
Assessment of Quality of Life (QoL) inequalities across clusters of European populations, countries, and healthcare systems, using EUonQoL-Kit questionnaires | At day 1
  Analysis of the QoL scores (dependent variable) according to individual-level variables as well as country/health system level variables (independent variables)
Socio-demographic and clinical factors potentially associated with QoL | At day 1
  Assessment of QoL disparities across different patient groups (by gender, ethnicity, religion, area, psychological and socio-economic factors, and education level)

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Brunelli, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
Locations (45):
- Mother Teresa University Hospital, Tirana, Albania
- Comprehensive Cancer Center, Vienna, Austria
- Kortrijk Kankercentrum AZ Groeninge, Kortrijk, Belgium
- Bulgarian Joint Cancer Network, Varna, Bulgaria
- Klinika za tumore Klinički bolnički centar Sestre milosrdnice, Zagreb, Croatia
- Cyprus Association of Cancer Patients and Friends (PASYKAF), Nicosia, Cyprus
- Masarykův onkologický ústav, Brno, Czechia
- Region Hovedstaden (Rigshospitalet), Hillerød, Denmark
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Sihtasutus Tartu Ülikooli Kliinikum, Tartu
- HUS Syöpäkeskus Helsingin Yliopistollinen Sairaala, Helsinki, Finland
- France (3):
  - lnstitut de Cancérologie de l'Ouest (ICO), Angers
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Petre Shotadze Tbilisi Medical Academy, Tbilisi, Georgia
- Germany (3):
  - Universitäres Centrum für Tumorerkrankungen (UCT), Frankfurt
  - Deutsches Krebsforschungszentrum (DKFZ), Heidelberg
  - Comprehensive Cancer Center Munich, Munich
- General Oncology Hospital of Athens - Saint Savvas, Athens, Greece
- Országos Onkológiai Intézet, Budapest, Hungary
- Trinity St. James's Cancer Institute, Dublin, Ireland
- Italy (4):
  - Istituto Tumori Giovanni Paolo II, IRCCS, Bari
  - Istituto Europeo di Oncologia, IRCCS, Milan
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Istituto Nazionale Tumori Regina Elena, Roma
- Riga East University Hospital, Riga, Latvia
- National Cancer Institute, Vilnius, Lithuania
- Oncologic Institute of Moldova, Chisinau, Moldova
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Oslo University Hospital (OUS), Oslo, Norway
- Poland (2):
  - Greater Poland Cancer Centre, Poznan
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy, Warsaw
- Instituto Português de Oncologia do Porto Francisco Gentil, E.P.E. (IPO-Porto), Porto, Portugal
- Romania (2):
  - Institutul Oncologic "Al. Trestioreanu" (IOB), Bucharest
  - The "Prof. Dr. Ion Chiricuta"Institute of Oncology (IOCN), Cluj-Napoca
- Oncology Institute of Vojvodina, Kamenitz, Serbia
- National Cancer Institute (Národný onkologický ústav), Bratislava, Slovakia
- Onkološki Inštitut Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Vall Hebron Institute of Oncology (VHIO), Barcelona
  - Fundación Instituto Valenciano de Oncología (IVO), Valencia
- Sweden (2):
  - Sahlgrenska comprehensive cancer centre, Gothenburg
  - Region Skåne - University Hospital Cancer Centre, Lund
- Turkey (Türkiye) (2):
  - Anadolu Medical Center, Gebze
  - Turkey Cancer Institute, Istanbul
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Anthoine E, Moret L, Regnault A, Sebille V, Hardouin JB. Sample size used to validate a scale: a review of publications on newly-developed patient reported outcomes measures. Health Qual Life Outcomes. 2014 Dec 9;12:176. doi: 10.1186/s12955-014-0176-2. PMID 25492701
- [Background] CAMPBELL DT, FISKE DW. Convergent and discriminant validation by the multitrait-multimethod matrix. Psychol Bull. 1959 Mar;56(2):81-105. No abstract available. PMID 13634291
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Kazis LE, Anderson JJ, Meenan RF. Effect sizes for interpreting changes in health status. Med Care. 1989 Mar;27(3 Suppl):S178-89. doi: 10.1097/00005650-198903001-00015. PMID 2646488
- [Background] de Haes JC, van Knippenberg FC, Neijt JP. Measuring psychological and physical distress in cancer patients: structure and application of the Rotterdam Symptom Checklist. Br J Cancer. 1990 Dec;62(6):1034-8. doi: 10.1038/bjc.1990.434. PMID 2257209
- [Background] Leyland AH, Groenewegen PP. Multilevel Modelling for Public Health and Health Services Research: Health in Context [Internet]. Cham (CH): Springer; 2020. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK565715/ PMID 33347097
- [Background] Liyanage H, Liaw ST, Jonnagaddala J, Hinton W, de Lusignan S. Common Data Models (CDMs) to Enhance International Big Data Analytics: A Diabetes Use Case to Compare Three CDMs. Stud Health Technol Inform. 2018;255:60-64. PMID 30306907
- [Background] Lyons MJ, Fernandez Poole S, Brownson RC, Lyn R. Place Is Power: Investing in Communities as a Systemic Leverage Point to Reduce Breast Cancer Disparities by Race. Int J Environ Res Public Health. 2022 Jan 6;19(2):632. doi: 10.3390/ijerph19020632. PMID 35055453
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN study reached international consensus on taxonomy, terminology, and definitions of measurement properties for health-related patient-reported outcomes. J Clin Epidemiol. 2010 Jul;63(7):737-45. doi: 10.1016/j.jclinepi.2010.02.006. PMID 20494804
- [Background] Petersen MA, Aaronson NK, Arraras JI, Chie WC, Conroy T, Costantini A, Dirven L, Fayers P, Gamper EM, Giesinger JM, Habets EJJ, Hammerlid E, Helbostad J, Hjermstad MJ, Holzner B, Johnson C, Kemmler G, King MT, Kaasa S, Loge JH, Reijneveld JC, Singer S, Taphoorn MJB, Thamsborg LH, Tomaszewski KA, Velikova G, Verdonck-de Leeuw IM, Young T, Groenvold M; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group. The EORTC CAT Core-The computer adaptive version of the EORTC QLQ-C30 questionnaire. Eur J Cancer. 2018 Sep;100:8-16. doi: 10.1016/j.ejca.2018.04.016. Epub 2018 Jun 21. PMID 29936066
- [Background] Reeve BB, Wyrwich KW, Wu AW, Velikova G, Terwee CB, Snyder CF, Schwartz C, Revicki DA, Moinpour CM, McLeod LD, Lyons JC, Lenderking WR, Hinds PS, Hays RD, Greenhalgh J, Gershon R, Feeny D, Fayers PM, Cella D, Brundage M, Ahmed S, Aaronson NK, Butt Z. ISOQOL recommends minimum standards for patient-reported outcome measures used in patient-centered outcomes and comparative effectiveness research. Qual Life Res. 2013 Oct;22(8):1889-905. doi: 10.1007/s11136-012-0344-y. Epub 2013 Jan 4. PMID 23288613
- [Background] Rock EP, Kennedy DL, Furness MH, Pierce WF, Pazdur R, Burke LB. Patient-reported outcomes supporting anticancer product approvals. J Clin Oncol. 2007 Nov 10;25(32):5094-9. doi: 10.1200/JCO.2007.11.3803. PMID 17991927
- [Background] Schag CA, Ganz PA, Heinrich RL. CAncer Rehabilitation Evaluation System--short form (CARES-SF). A cancer specific rehabilitation and quality of life instrument. Cancer. 1991 Sep 15;68(6):1406-13. doi: 10.1002/1097-0142(19910915)68:63.0.co;2-2. PMID 1873793
- [Background] Schipper H, Clinch J, McMurray A, Levitt M. Measuring the quality of life of cancer patients: the Functional Living Index-Cancer: development and validation. J Clin Oncol. 1984 May;2(5):472-83. doi: 10.1200/JCO.1984.2.5.472. PMID 6374052
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Epidemiology. 2007 Nov;18(6):800-4. doi: 10.1097/EDE.0b013e3181577654. PMID 18049194
- [Background] Wainer H. (2000). Computerized Adaptive testing: A Primer (2nd ed.). Mahwah, New Jersey: Lawrence Erlbaum Associates, Inc.
- [Background] Velikova G, Coens C, Efficace F, et al. Health-related quality of life in EORTC clinical trials - 30 years of progress from methodological developments to making a real impact on oncology practice. EJC Suppl 2012;10(1):141-9.
- [Background] Petersen MA, Groenvold M, Bjorner JB, Aaronson N, Conroy T, Cull A, Fayers P, Hjermstad M, Sprangers M, Sullivan M; European Organisation for Research and Treatment of Cancer Quality of Life Group. Use of differential item functioning analysis to assess the equivalence of translations of a questionnaire. Qual Life Res. 2003 Jun;12(4):373-85. doi: 10.1023/a:1023488915557. PMID 12797710
- [Background] Cronbach LJ. Coefficient alpha and the internal structure of tests. Psychometrika 1951;16(3):297-334.
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Derived] Apolone G, Costantini M, Caselli L, Bos N, Caraceni A, Ciliberto G, Couespel N, Ferrer M, Groenvold M, Kaasa S, Lombardo C, Pietrobon R, Pravettoni G, Sirven A, Vachon H, Velikova G, Garin O, Gilbert A, Machiavelli A, Marzorati C, Miceli R, Pe M, Petersen MA, Tanzilli A, van Schelven F, Dantas C, Minnee-van Braak I, Pinnavaia L, Brunelli C. Validation of the European Oncology toolkit for the self-assessment of Quality of Life (EUonQoL-Kit) in cancer patients and survivors: study protocol of a pan European survey. BMC Public Health. 2024 Dec 18;24(1):3517. doi: 10.1186/s12889-024-21008-4. PMID 39696103